CLINICAL TRIAL: NCT03435614
Title: Signs and Symptoms of Opioid-associated Iatrogenic Withdrawal in Critically Ill Adults
Acronym: SOWA-ICU
Status: Completed | Type: Observational
Sponsor: Marc M. Perreault (Other)
Responsible Party: Sponsor-Investigator, Marc M. Perreault, Pharmacist, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Other Study IDs: 2018-4305
Record Dates: First submitted 2018-02-09; First posted 2018-02-19 (Actual); Results first posted 2021-01-28 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Substance Withdrawal Syndrome
Keywords: Opioid; Withdrawal; Critically ill adults; Cortisol
MeSH Terms: conditions — Substance Withdrawal Syndrome | interventions — Analgesics, Opioid; Analgesics; Narcotics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically ill patients: Mechanically ventilated critically ill adults receiving regular opioids for more than 72 hours will be prospectively followed for the emergence of withdrawal symptoms upon weaning of opioids.
  Interventions: Drug: Opioids

INTERVENTIONS:
Drug: Opioids — Once an opioid dose reduction of 10% or greater is achieved, a daily assessment will be conducted by a physician using the DSM-5 criteria for opioid withdrawal. In addition, signs and symptoms of withdrawal will be collected daily by a blinded investigator.
  Other Names: Analgesics; Narcotics

SUMMARY:
Mechanically ventilated critically ill adults may require prolonged administration of opioids to facilitate ventilator support and maintain comfort. The prolonged use has been associated with withdrawal symptoms upon rapid weaning in critically ill patients, known as the opioid-associated withdrawal syndrome (OIWS). Such withdrawal symptoms are well described in the paediatric population, however there is a lack of information in the adult population. Currently there is no bedside tool to rapidly identify such patients. Recognition of withdrawal symptoms is the basis for the development of an assessment tool to identify patients with OIWS.

DETAILED DESCRIPTION:
Objectives:

1. To identify specific signs and symptoms of OIWS in mechanically ventilated adult intensive care unit (ICU) patients receiving at least 72 hours of regular opioids at the Montreal General Hospital (MGH) and the Royal Victoria Hospital (RVH) from February to October 2018.
2. To determine if a change in serum cortisol is associated with the presence of OIWS.

Hypotheses:

1. Considering our first objective is purely descriptive, no hypothesis can be stated.
2. OIWS is associated with an increase in serum cortisol.

Methods:

A prospective multicentre observational study will be carried out in two university-affiliated hospital ICUs (Montreal General Hospital and Royal Victoria Hospital). All mechanically ventilated adult ICU patients receiving regular (continuous or intermittent) opioids for more than 72 hours will be prospectively screened daily for withdrawal symptoms once the opioid dose is reduced by 10% or more. From that moment, daily evaluation by a physician using the Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) criteria for opioid withdrawal will be conducted. Concomitantly, signs and symptoms of withdrawal will be collected by an investigator blinded to the DSM-5 assessment. These assessments will continue daily until the patient is transferred out of ICU or a maximum of 14 days and will be repeated once more between day 1 and day 4 post-transfer out of ICU.

A serum cortisol will be drawn on the first day of dose reduction by 10% or more (baseline) and will be repeated either after 72 hours or upon patient discharge from the ICU, whichever one occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring mechanical ventilation and receiving continuous or regular intermittent opioids for at least 72 hours.
* Weaning of at least 10% from previous stable opioid dose. A weaning episode is defined as a ≥ 10% decrease in the total stable opioid dose received over 4 hours for opioid infusions and over 12 hours for intermittent opioid administration.

Exclusion Criteria:

* Patient for whom consent cannot be obtained
* Patient and/or family unable to communicate in French or English
* Patient who is deaf without appropriate hearing aid
* Imminent and predictable death (< 72 hours) according to medical team
* Severe brain injury, defined as Glasgow Coma Scale (GCS) score of 8 or less at ICU admission
* Moderate brain injury, defined as GCS between 9 and 12, with elevated intracranial pressure (ICP > 20 mmHg) which requires ICP monitoring and osmotherapy
* Acute neurological condition (e.g. status epilepticus, encephalopathy, stroke). If the acute neurological condition resolves within 72 hours, the patient may be included in the study.
* Substance abuse prior to ICU admission.

  * Chronic alcohol use defined as alcohol consumption of more than 2 drinks/day and/or more than 14 drinks/week for men and 9 drinks/week for women.
  * Chronic use of illicit drugs and amphetamines (except amphetamines taken for therapeutic purposes) defined as a consumption of at least 3 times per week.
  * Chronic use of opioids (e.g. transdermal fentanyl, methadone, hydromorphone, etc.) defined as a consumption of at least 3 times per week.
* Readmission to the MGH or RVH ICU during the recruitment period (limit of one study entry per patient)
* Spinal cord injury above the lumbar region

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated adult ICU patients receiving continuous or regular intermittent opioids for more than 72 hours.
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Soleil Delisle, MSc, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Marc M Perreault, PharmD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Marc-Alexandre Duceppe, MSc, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chiu AW, Contreras S, Mehta S, Korman J, Perreault MM, Williamson DR, Burry LD. Iatrogenic Opioid Withdrawal in Critically Ill Patients: A Review of Assessment Tools and Management. Ann Pharmacother. 2017 Dec;51(12):1099-1111. doi: 10.1177/1060028017724538. Epub 2017 Aug 9. PMID 28793780
- [Background] Wang PP, Huang E, Feng X, Bray CA, Perreault MM, Rico P, Bellemare P, Murgoi P, Gelinas C, Lecavalier A, Jayaraman D, Frenette AJ, Williamson D. Opioid-associated iatrogenic withdrawal in critically ill adult patients: a multicenter prospective observational study. Ann Intensive Care. 2017 Sep 2;7(1):88. doi: 10.1186/s13613-017-0310-5. PMID 28866754
- [Background] Cammarano WB, Pittet JF, Weitz S, Schlobohm RM, Marks JD. Acute withdrawal syndrome related to the administration of analgesic and sedative medications in adult intensive care unit patients. Crit Care Med. 1998 Apr;26(4):676-84. doi: 10.1097/00003246-199804000-00015. PMID 9559604

RESULTS

PARTICIPANT FLOW:
Groups:
- Iatrogenic Withdrawal Syndrome (IWS) Positive: Group of patients displaying signs and symptoms of IWS
- Iatrogenic Withdrawal Syndrome (IWS) Negative: Group of patients not displaying signs and symptoms of IWS
Period: Overall Study
Arm/Group | Iatrogenic Withdrawal Syndrome (IWS) Positive | Iatrogenic Withdrawal Syndrome (IWS) Negative
Started | 6 | 23
Completed | 6 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 1128 patients screened; 59 eligible as per entry criteria; 29 enrolled and included in the analysis
Groups:
- Opioid Iatrogenic WIthdrawal Syndrome (OIWS) Positive Patients: Mechanically ventilated critically ill adults receiving regular opioids for more than 72 hours whose at least one daily DSM-5 assessment for OIWS was positive following the reduction in opioid dose (opioid dose reduction of 10% or greater).
- Opioid Iatrogenic Withdrawal Syndrome (OIWS) Negative Patients: Mechanically ventilated critically ill adults receiving regular opioids for more than 72 hours whose daily DSM-5 assessments for OIWS remained negative for the duration of follow up following the reduction in opioid dose (opioid dose reduction of 10% or greater).
- Total: Total of all reporting groups
Arm/Group | Opioid Iatrogenic WIthdrawal Syndrome (OIWS) Positive Patients | Opioid Iatrogenic Withdrawal Syndrome (OIWS) Negative Patients | Total
Number analyzed (Participants) | 6 | 23 | 29
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 70 [62.0 to 77.3] | 64 [44.0 to 74.0] | 65 [47.5 to 75.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 8
  Male | 4 | 17 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 6 | 17 | 23
  Hispanic | 0 | 2 | 2
  Black | 0 | 2 | 2
  MIddle Eastern | 0 | 2 | 2
Serum Creatinine at ICU admission (umol/L) [Median (Inter-Quartile Range); unit: umol/L] | 124 [78 to 307] | 136 [71 to 223] | 132 [74 to 222]
Reason for ICU admission (ICD-10) [Count of Participants; unit: Participants]
  Diseases of the circulatory system | 1 | 6 | 7
  External causes of morbidity and mortality (trauma) | 1 | 5 | 6
  Infectious and parasitic diseases | 0 | 5 | 5
  Diseases of the digestive system | 3 | 2 | 5
  Diseases of the respiratory system | 0 | 4 | 4
  Other | 1 | 1 | 2
Length of ICU stay [Median (Inter-Quartile Range); unit: Days] | 16.5 [9.5 to 38.0] | 16 [9.0 to 34.0] | 16.0 [9.0 to 35.0]
Duration of mechanical ventilation [Median (Inter-Quartile Range); unit: Days] | 9.0 [7.3 to 37.3] | 9.0 [5.0 to 26.0] | 9.0 [5.5 to 27.0]
Co-morbidities [Number; unit: participants]
  Hypertension | 3 | 12 | 15
  Coronary artery disease | 2 | 11 | 13
  Diabetes | 1 | 8 | 9
  Chronic kidney disease | 1 | 5 | 6
  Chronic obstructive pulmonary disease | 2 | 4 | 6
  Other | 3 | 9 | 12
As needed use of opioids prior to ICU admission [Count of Participants; unit: Participants] | 0 | 1 | 1
Use of benzodiazepines prior to ICU admission [Count of Participants; unit: Participants] | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Description of Signs and Symptoms of OIWS in Patients Who Scored Positive for Withdrawal Syndrome (OIWS) According to Diagnostic and Statistical Manual of Mental Disorders (DSM-5) Criteria
Description: Percentage of daily assessments associated with each of the following signs and symptoms experienced by patients with and without OIWS (Restlessness (Richmond Agitation-Sedation scale = 1), Agitation (RASS > 1), Anxiety, Hallucinations, Insomnia/sleep disturbance (< 4 hours of continuous sleep), Mydriasis (Pupil diameter > 2 mm) and systolic blood pressure (SBP) > 140 mmHg. These assessments were performed once daily.
  Note that for the group of patients experiencing IWS, the data on signs and symptoms are limited to the assessment on the day that patients experienced OIWS.
  The signs and symptoms presented (Restlessness; Agitation; Anxiety, Hallucinations, Insomnia/sleep disturbance; mydriasis; SBP > 140) were selected based on a > 15 % absolute difference between both groups which was judged to be clinically significant.
Time Frame: From first day of opioid dose reduction until transfer out of Intensive care unit (ICU) or a maximum of 14 days, including one further assessment post-ICU transfer
Measure: Number; unit: percentage of assessments
Groups:
- IWS Positive: Group of patients with OIWS positive as per DSM-V criteria
- IWS Negative: Group of patients without OIWS as per DSM-V criteria
Arm/Group | IWS Positive | IWS Negative
Number analyzed (Participants) | 6 | 23
percentage of assessments
  Restlessness (RASS = 1) | 28.6 | 13.6
  Agitation (RASS > 1) | 28.6 | 4.9
  Anxiety | 57.1 | 30.6
  Hallucinations | 28.6 | 11.2
  Insomnia/Sleep disturbance (< 4 hours of continuous sleep) | 66.7 | 21.4
  Mydriasis (pupil size > 2mm) | 100 | 77.8
  Systolic Blood Pressure (SBP) > 140 mmHg | 85.7 | 53
Statistical Analysis 1: Comparison: IWS Positive vs IWS Negative; Test type: Other; We selected the individual signs and symptoms associated with the presence of OIWS based on a difference of greater than 15 % in the assessments between the group with OIWS and the group not displaying OIWS. This 15 % difference was judged to be of clinical significance. The signs and symptoms which did not meet this difference were not considered (data not available)

2. Secondary Outcome: Change in Serum Cortisol Level
Description: Cortisol level were drawn on the first day of opioid weaning and repeated 72 hours after onset of weaning
Time Frame: Baseline cortisol on first day of opioid dose reduction and on day 3 post-dose reduction, or on day of transfer out of ICU if patient is transferred before day 3.
Population: Only 9 patients had two sets of blood samples drawn for cortisol levels measurement
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | IWS Positive | IWS Negative
Number analyzed (Participants) | 1 | 8
nmol/L | -146 | -37 [-62 to 93]

ADVERSE EVENTS:
Time Frame: Symptom assessments were collected daily until transfer out of ICU, death or 14 days after start of patient remained in ICU; If patient was transferred, one additional data was collected up to 96 hours post-transfer out of ICU
Description: Observational study of IWS - Non interventional
Arm/Group | Critically Ill Patients
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-04): https://cdn.clinicaltrials.gov/large-docs/14/NCT03435614/Prot_SAP_000.pdf